Predictors of Speech Ability in Down Syndrome Statistical Analysis Plan NCT05016037 April 24, 2025

## Statistical Analysis Plan

There are three levels of analysis that were completed. The first included descriptive statistics for means and standard deviations for study dependent measures (e.g., speech accuracy scores on standardized tests). The second level included testing for pre- versus post differences on key dependent measures using repeated measures means tests as appropriate (e.g., paired sample t tests). The third and final level included completing correlational analysis to explore relationships among the pre post gain scores and dependent measures such as expressive vocabulary level, receptive language level and age level.